CLINICAL TRIAL: NCT00337168
Title: A Phase II Trial of Cytarabine and Clofarabine in Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: S0530 Cytarabine and Clofarabine in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0530; U10CA032102 (NIH); SWOG-S0530 (Other: SWOG)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induc, ReInduc, Consol, clofarabine, cytarabine (Experimental): Induction: 40mg/m2/d; IV over 1 hr; days 1-5 Re-induction (if necessary): 40mg/m2/d; IV over 1 hr; days 1-5 Consolidation: 40mg/m2/d; IV over 1 hr; days 1-4
  Interventions: Drug: clofarabine; Drug: cytarabine

INTERVENTIONS:
Drug: clofarabine — Induction: 40mg/m2/d; IV over 1 hr; days 1-5 Re-induction (if necessary): 40mg/m2/d; IV over 1 hr; days 1-5 Consolidation: 40mg/m2/d; IV over 1 hr; days 1-4
Drug: cytarabine — Induction: 1g/m2/d; IV over 2 hrs; days 1-5 Re-induction (if necessary): 1g/m2/d; IV over 2 hrs; days 1-5 Consolidation: 1g/m2/d; IV over 2 hrs; days 1-4

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving cytarabine together with clofarabine works in treating patients with relapsed or refractory acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Primary objective:

* Determine whether the complete remission rate in adult patients with relapsed or refractory acute lymphoblastic leukemia (ALL) is sufficiently high after treatment with cytarabine and clofarabine to warrant further investigation.

Secondary objectives:

* Estimate the frequency and severity of toxicities associated with this dosing schedule of cytarabine and clofarabine.
* Investigate, preliminarily, the prognostic effects of cytogenetic features on response to treatment in these patients.

Other objectives (if funding allows):

* Investigate, preliminarily, the prognostic effects of laboratory correlates (expression of nucleoside transporters, expression of other pertinent genes by tissue microarray) and FISH features on response to treatment in these patients

OUTLINE: This is an open-label, multicenter study.

* Induction therapy (1 or 2 courses): Patients receive induction therapy comprising clofarabine IV over 1 hour followed 4 hours later by cytarabine IV over 2 hours on days 1-5 (course 1). Patients who achieve a response (5-25% blasts in the bone marrow with a ≥ 50% reduction in blasts from initial bone marrow aspirate) receive 1 more course of induction therapy beginning no later than day 45. Patients who achieve complete remission (< 5% blasts in the bone marrow) after 1 or 2 courses of induction therapy may proceed to consolidation therapy.
* Consolidation therapy (1 course): Beginning within 60 days after the first day of the last induction therapy, patients may receive consolidation therapy comprising clofarabine IV over 1 hour followed 4 hours later by cytarabine IV over 2 hours on days 1-4.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior morphologic diagnosis of acute lymphoblastic leukemia (ALL)

  * No M0, mixed lineage, or L3 (Burkitt's) ALL
* Refractory to a standard induction regimen OR relapsed after successful prior induction therapy

  * Standard induction regimen is defined as any program of treatment that includes vincristine and prednisone or high-dose cytarabine/mitoxantrone
  * Any number of inductions or remissions allowed
* Must have evidence of ALL in bone marrow or peripheral blood

  * Immunophenotyping of the blood or bone marrow lymphoblasts must be performed to determine lineage (B cell, T cell, or mixed B/T cell)
  * No extramedullary only disease in the absence of bone marrow or blood involvement
  * Co-expression of myeloid antigens (CD13 and CD33) allowed
* Patients with Philadelphia chromosome-positive (Ph+) ALL or bcr/abl-positive ALL who were previously eligible for imatinib mesylate treatment must have received imatinib mesylate either alone or in combination with chemotherapy for ALL and must have either failed treatment or been unable to tolerate treatment
* No CNS involvement as determined by lumbar puncture (for previous CNS history or clinical signs or symptoms of CNS) or by clinical exam (if no previous history or signs/symptoms)
* Must be registered on SWOG-S9910 and SWOG-9007

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 1.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* No psychiatric disorders that would interfere with study compliance
* No uncontrolled systemic fungal, bacterial, viral, or other infection
* No other severe concurrent disease
* No other serious or poorly controlled medical condition that would preclude study participation
* No history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing motor or sensory neuropathy ≥ grade 2
* No other prior malignancies, except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer in complete remission
  * Any other prior cancer for which the patient has been disease free for ≥ 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior clofarabine
* More than 2 weeks since prior chemotherapy, major surgery, or other investigational agents
* More than 6 weeks since prior monoclonal antibodies
* Prior allogeneic or autologous bone marrow transplant allowed provided the following criteria are met:

  * More than 90 days since transplant
  * No acute graft-versus-host disease (GVHD) ≥ grade 2 OR moderate or severe limited chronic GVHD OR extensive chronic GVHD of any severity
* Prior maintenance therapy with steroids, vincristine, and/or anti-metabolite agents, such as, but not limited to, mercaptopurine, thioguanine, or methotrexate allowed
* Concurrent hydroxyurea allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, MD, Study Chair — The Cleveland Clinic; Jerry Radich, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (91):
- United States (91):
  - Providence Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Stanford Cancer Center, Stanford, California
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Frontier Cancer Center, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction: Clofarabine (40 mg per meters squared per day) and cytarabine (1 g per meters squared per day)
Period: Overall Study
Arm/Group | Induction
Started | 37
Eligible | 37
Eligible and Treated | 36
Completed | 29
Not Completed | 8
Not completed — Death | 5
Not completed — Not protocol specified | 2
Not completed — Did not start therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Induction
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 41 [20 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Remission
Description: Complete remission is defined as: less than 5% bone marrow blasts, neutrophils greater or equal to 1,000 per microliter, platelets greater than 100,000 per microliter, no blasts in the peripheral blood, and no extramedullary disease
Time Frame: Between day 28 and day 35 inclusive
Population: Eligible patients who started therapy
Measure: Number; unit: participants
Arm/Group | Induction
Number analyzed (Participants) | 36
participants | 3

2. Secondary Outcome: Expression of Nucleoside Transporters
Description: Expression was examined in paraffin-embedded tissue by immunohistochemistry. Intensities were scored on a 0-2+ scale. High expression was a score of 2+.
Time Frame: On average, two weeks before treatment started
Population: Eligible patients who submitted paraffin-embedded tissue
Measure: Number; unit: participants
Arm/Group | Induction
Number analyzed (Participants) | 13
participants
  High expression of hENT1 | 7
  High expression of hCNT3 | 6
  High expression of dCK cytoplasmic | 4
  High expression of dCK nuclear | 4

3. Secondary Outcome: Number of Patients With Very Poor Risk Cytogenetics
Time Frame: On average, 2 weeks before treatment started
Population: Eligible patients with acceptable centrally reviewed cytogenetics
Measure: Number; unit: participants
Arm/Group | Induction
Number analyzed (Participants) | 17
participants | 10

4. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: Patients were assess for adverse events after each induction cycle (up to two cycles) and after the one consolidation cycle
Population: Eligible patients who started therapy
Measure: Number; unit: Participants with a given type of AE
Groups:
- Induction: Up to two induction cycles with clofarabine and cytarabine
Arm/Group | Induction
Number analyzed (Participants) | 36
Participants with a given type of AE
  ALT, SGPT (serum glutamic pyruvic transaminase) | 5
  AST, SGOT (serum glut oxaloacetic transaminase) | 7
  Albumin, serum-low (hypoalbuminemia) | 3
  Anorexia | 1
  Ascites (non-malignant) | 2
  Bilirubin (hyperbilirubinemia) | 3
  Calcium, serum-low (hypocalcemia) | 1
  Colitis | 1
  Colitis, infectious (e.g., Clostridium difficile) | 2
  Confusion | 1
  Creatinine | 4
  DIC (disseminated intravascular coagulation) | 1
  Death not assoc with CTCAE term-Multi-organ fail | 1
  Dermatology/Skin-Other (Specify) | 1
  Diarrhea | 2
  Dyspnea (shortness of breath) | 1
  Edema: limb | 1
  Fatigue (asthenia, lethargy, malaise) | 2
  Febrile neutropenia | 14
  Glucose, serum-high (hyperglycemia) | 1
  Hemoglobin | 13
  Hypotension | 3
  Hypoxia | 1
  INR | 1
  Infec with Gr 3\4 neutrophils - Bladder (urin | 1
  IInfec with Gr 3\4 neutrophils - Blood | 9
  Infec with Gr 3\4 neutrophils - Catheter-rela | 1
  Infec with Gr 3\4 neutrophils - Colon | 2
  Infec with Gr 3\4 neutrophils - Conjunctiva | 1
  Infec with Gr 3\4 neutrophils - Larynx | 1
  Infec with Gr 3\4 neutrophils - Lung (pneumon | 2
  Infec with Gr 3\4 neutrophils - Skin (celluli | 1
  Infec with Gr 3\4 neutrophils - Urinary tract | 1
  Infec with Gr 3\4 neutrophils - Wound | 1
  Infection with unknown ANC - Lung (pneumonia) | 1
  Infection-Other (Specify) | 1
  Leukocytes (total WBC) | 11
  Liver dysfunction/failure (clinical) | 1
  Lymphopenia | 7
  Mental status | 1
  Neutrophils/granulocytes (ANC/AGC) | 18
  PTT (Partial thromboplastin time) | 1
  Pain - Abdomen NOS | 1
  Pain - Back | 1
  Pain - Bone | 1
  Platelets | 20
  Pleural effusion (non-malignant) | 1
  Pneumonitis/pulmonary infiltrates | 1
  Potassium, serum-high (hyperkalemia) | 1
  Potassium, serum-low (hypokalemia) | 4
  Pruritus/itching | 1
  Renal failure | 3
  Restrictive cardiomyopathy | 1
  Sodium, serum-high (hypernatremia) | 1
  Sodium, serum-low (hyponatremia) | 2
  Supraventricular and nodal arrhythmia | 1
  Tumor lysis syndrome | 1
  Typhlitis (cecal inflammation) | 1
  Uric acid, serum-high (hyperuricemia) | 1

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported
Description: Regular investigator assessments are reported after each cycle of protocol treatment
Arm/Group | Induction
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (N=36)
Febrile neutropenia (Blood and lymphatic system disorders) | 14
Hemoglobin (Blood and lymphatic system disorders) | 18
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 3
Ascites (non-malignant) (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 11
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Pain - Abdomen NOS (Gastrointestinal disorders) | 6
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Edema: limb (General disorders) | 6
Fatigue (asthenia, lethargy, malaise) (General disorders) | 10
Rigors/chills (General disorders) | 3
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 9
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Colon (Infections and infestations) | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 11
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 11
Alkaline phosphatase (Investigations) | 5
Bilirubin (hyperbilirubinemia) (Investigations) | 10
Creatinine (Investigations) | 7
INR (International Normalized Ratio of prothrombin time) (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 11
Lymphopenia (Investigations) | 7
Metabolic/Laboratory-Other (Specify) (Investigations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 18
PTT (Partial thromboplastin time) (Investigations) | 3
Platelets (Investigations) | 20
Weight loss (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 5
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 9
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5
Pain - Back (Musculoskeletal and connective tissue disorders) | 3
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3
Pain - Head/headache (Nervous system disorders) | 10
Confusion (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 4
Mood alteration - depression (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 4
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No